CLINICAL TRIAL: NCT07173673
Title: A Prospective, Multi-center, Randomized Clinical Trial to Evaluate the Detection of Atrial Fibrillation Using Artificial Intelligence-Enhanced Electrocardiography (SmartECG-AFrisk) Compared With Usual Care in Patients With Suspected Atrial Fibrillation: DEEP-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2024-0069
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (General Practice) (Active Comparator): Symptom-based evaluation by physicians, including 12-lead ECG, Holter monitoring, or patch ECG at least once within 6 months
  Interventions: Other: Usual Care (General Practice)
- AI-ECG Guided Care (SmartECG-AFrisk) (Experimental): Monitoring strategy determined by SmartECG-AFrisk risk score (≥50 = high-risk vs <50 = low-risk).
  Interventions: Device: AI-ECG Guided Care (SmartECG-AFrisk)

INTERVENTIONS:
Other: Usual Care (General Practice) — Participants receive routine care based on current clinical guidelines. Symptom-driven evaluation is performed by physicians, including at least one diagnostic test within 6 months such as a standard 12-lead ECG, Holter monitoring, or patch ECG. The choice and frequency of monitoring are determined by physician discretion, reflecting real-world practice patterns.
  Arms: Usual Care (General Practice)
Device: AI-ECG Guided Care (SmartECG-AFrisk) — Participants undergo SmartECG-AFrisk analysis of baseline 12-lead ECGs recorded in sinus rhythm. The algorithm calculates an atrial fibrillation risk score, classifying participants as high-risk (score ≥50) or low-risk (<50). Monitoring strategies are adapted accordingly: high-risk participants undergo targeted and potentially repeated ECG monitoring using 12-lead ECG, Holter, or patch ECG, while low-risk participants follow standard guideline-based care.
  Arms: AI-ECG Guided Care (SmartECG-AFrisk)

SUMMARY:
"The DEEP-AF study is a prospective, multi-center, randomized clinical trial evaluating the effectiveness of an artificial intelligence-enhanced electrocardiography algorithm (SmartECG-AFrisk) for early detection of atrial fibrillation (AF) in adults with suspected AF but no prior diagnosis. A total of 1,230 participants will be enrolled across 13 centers in Korea and randomized 1:1 into standard care or AI-guided care arms.

In the standard care arm, diagnostic evaluation follows clinical guidelines with symptom-based use of 12-lead ECG, Holter, or patch ECG. In the AI-guided arm, baseline 12-lead ECGs are analyzed using SmartECG-AFrisk to calculate an AF risk score. Participants are classified as high-risk (score ≥50) or low-risk (<50), and monitoring strategies are determined accordingly, enabling targeted ECG monitoring for high-risk individuals.

The primary objective is to compare the 6-month incidence of newly diagnosed AF between the two arms. Secondary endpoints include AF detection differences between risk groups, healthcare resource utilization per AF diagnosis, anticoagulation initiation rates, major clinical events (stroke, embolism, bleeding, mortality), and patient satisfaction.

This study aims to demonstrate whether integrating AI-driven ECG risk stratification into routine care improves AF detection and optimizes healthcare resource use in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Adults ≥30 years old

* - Symptoms suggestive of atrial fibrillation (palpitations, dizziness, syncope, dyspnea, chest discomfort)
* - No evidence of AF on baseline 12-lead ECG
* - No prior history of AF diagnosis

Exclusion Criteria:

* - Prior diagnosis of atrial fibrillation
* - Life expectancy ≤ 1 year

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1230 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
New diagnosis of atrial fibrillation within 6 months. (confirmed by ECG, Holter, or patch ECG) | Baseline (randomization) to 6 months after enrollment. Event date is defined as the first ECG/Holter/patch ECG documenting AF during the 6-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No